CLINICAL TRIAL: NCT02152592
Title: Controlled-Release Oxycodone Versus Naproxen at Home After Ambulatory Surgery: A Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Bjorn Stessel, MD, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11524; 2006-003545-17 (EudraCT Number)
Record Dates: First submitted 2014-05-28; First posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Postoperative Pain After Ambulatory Surgery
Keywords: Postoperative pain; Ambulatory surgery; NSAIDS; CR Oxycodone; Compliance to study medication
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PCM/NAPR group (No Intervention): paracetamol 1000 mg orally four times a day for 48 hours postoperatively and naproxen 500 mg orally twice a day for 48 hours postoperatively (standard hospital pain protocol for treatment of acute postoperative pain at home after painful day-case surgery)
- PCM/Oxy1 group (Active Comparator): Controlled Release oxycodone 10 mg orally twice a day for 24 hours and paracetamol 1000 mg orally four times a day for 48 hours postoperatively
  Interventions: Drug: PCM/Oxy1
- PCM/Oxy2 group (Active Comparator): CR oxycodone 10 mg orally twice a day for 48 hours and paracetamol 1000 mg orally four times a day for 48 hours postoperatively
  Interventions: Drug: PCM/Oxy2

INTERVENTIONS:
Drug: PCM/Oxy1 — Controlled Release oxycodone 10 mg orally twice a day for 24 hours
  Arms: PCM/Oxy1 group
Drug: PCM/Oxy2 — CR oxycodone 10 mg orally twice a day for 48 hours
  Arms: PCM/Oxy2 group

SUMMARY:
the primary objective of this study is to assess and compare the efficacy, safety and benefits of Controlled Release (CR) oxycodone/paracetamol with our current pain protocol (paracetamol/naproxen) in the treatment of acute postoperative pain at home after painful day-case surgery. We hypothesize that ambulatory patients postoperatively treated with oxycodone/paracetamol will achieve better pain relief with equal side effects compared to patients treated with paracetamol/naproxen.

Our second goal is to assess analgesic adherence in the outpatient setting.

Endpoints:

Primary endpoints: pain intensity (Visual analogue scale) Secondary endpoints: - side-effects/ adverse effects of study medication

* patient satisfaction with pain treatment
* compliance to study medication

Study design:

Patients scheduled for painful ambulatory surgery (knee arthroscopy, unilateral open or laparoscopic inguinal hernia repair) will be enrolled in an open randomized controlled trial (RCT) at our pre-assessment clinic.

Subjects will be enrolled by a study nurse and will be randomized into one of three study treatment groups using a computer-generated list. Patients in group 1 (PCM/NAPR) are assigned to postoperative analgesia using naproxen 500 mg orally twice a day for 48 hours postoperatively. Patients assigned to group 2 (PCM/Oxy1) receive CR oxycodone 10 mg orally twice a day for 24 hours. Patients in group 3 (PCM/Oxy2) are postoperatively treated witch CR oxycodone 10 mg orally twice a day for 48 hours. All patients also receive paracetamol 1000 mg orally four times a day for 48 hours postoperatively.

Recovery after discharge will be assessed using a diary for up to 48 hours after surgery. Three times a day, patients have to rate pain at rest and movement (VAS), fatigue, nausea, vomiting, pruritus, miction problems, pyrosis, and abdominal complaints. Furthermore, compliance to the use of the study medication will be assessed by checking whether the patients took the study medication as prescribed and if any other pain medication was used. Compliance will be assessed three times a day and patients will be divided into three groups according to medication use: always = full compliance, sometimes = partial compliance, or never = no compliance.

Finally, overall satisfaction with the postoperative pain treatment will be assessed (score 0-10).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for painful ambulatory surgery (knee arthroscopy, unilateral open or laparoscopic inguinal hernia repair)
* American Society of Anesthesiologists (ASA) physical classification I or II

Exclusion Criteria:

* cognitive impairment,
* preoperative pharmacologic pain treatment
* allergy to or a contraindication for taking the study medication (e.g. paracetamol, oxycodone, naproxen or another NSAID)
* porphyria
* pregnancy or lactation
* history of severe renal, hepatic, pulmonary, or cardiac failure
* current symptoms or history of gastrointestinal bleeding, ileus or chronic obstipation
* history of substance abuse, or use of medication with a suppressive effect on the central nervous system

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
a difference on a pain visual analogue scale between study groups | up to 48 hours
  a difference of 15mm or more on a visual analogue scale between three study groups is considered clinically relevant

SECONDARY OUTCOMES:
Incidence of adverse effects of study medication | up to 48 hours

OTHER OUTCOMES:
Adherence to study medication | up to 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Maastricht University Medical Center+, The Netherlands, Maastricht, Netherlands

REFERENCES:
- [Derived] Stessel B, Theunissen M, Fiddelers AA, Joosten EA, Kessels AG, Gramke HF, Marcus MA. Controlled-release oxycodone versus naproxen at home after ambulatory surgery: a randomized controlled trial. Curr Ther Res Clin Exp. 2014 Nov 28;76:120-5. doi: 10.1016/j.curtheres.2014.10.001. eCollection 2014 Dec. PMID 25516773